CLINICAL TRIAL: NCT04241705
Title: Evaluation of the Effect of Targeted Mass Drug Administration and Reactive Case Detection on Malaria Transmission and Elimination in East Hararghe Zone, Oromia, Ethiopia
Brief Title: Evaluation of Targeted Mass Drug Administration for Malaria in Ethiopia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Armauer Hansen Research Institute, Ethiopia (Other)
Collaborators: Addis Continental Institute of Public Health (Other); U.S. President's Malaria Initiative (Unknown); U.S. Centers for Disease Control and Prevention (Unknown); United States Agency for International Development (USAID) (U.S. Federal Agency); Ethiopian Federal Ministry of Health (Unknown); Oromia Regional Health Bureau (Unknown); Tulane University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1
Record Dates: First submitted 2020-01-02; First posted 2020-01-27 (Actual); Last update posted 2020-06-12 (Actual); Status verified 2020-06

CONDITIONS: Malaria
Keywords: Targeted mass drug administration; Reactive case detection
MeSH Terms: conditions — Malaria | interventions — Artemether, Lumefantrine Drug Combination; Primaquine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control arm (Active Comparator): The control arm will provide optimized malaria control interventions that includes strengthened surveillance systems and commodities management, scale-up of vector control and case management services.
  Interventions: Other: Optimized malaria control interventions
- Reactive Case Detection (RCD) arm (Active Comparator): Optimized malaria control interventions as in the control arm. In addition, following identification of microscopy or RDT positive, passively-detected index cases at the health post or health center; individuals who reside within a 100-meter radius of the index case will receive diagnosis for malaria using a conventional RDT. Positive individuals will receive treatment and follow-up as per the national treatment guidelines. 14 days of primaquine (PQ) will only be administered to those found to be normal upon G6PD testing. Additional procedures will include the collection of a dried blood spot.
  Interventions: Other: Treatment of positive individuals per national treatment guidelines; Other: Optimized malaria control interventions
- Targeted Mass Drug Administration (tMDA) arm (Experimental): Optimized malaria control interventions as in the control arm. In addition, following identification of microscopy or RDT positive index cases at the health post or health center, all eligible individuals who reside within a 100-meter radius of the index case will receive presumptive treatment with artemether-lumefantrine (AL) plus 14 days of primaquine (PQ) (0.25mg/kg daily). 14 days of primaquine (PQ) will only be administered to those found to be normal upon G6PD testing.
  Interventions: Other: Presumptive treatment with artemether-lumefantrine (AL) plus 14 days of primaquine (PQ); Other: Optimized malaria control interventions

INTERVENTIONS:
Other: Treatment of positive individuals per national treatment guidelines — Treatment for everyone except children <6 months of age, pregnant women, women breastfeeding children <6 months of age, and women 12-49 years of age with an unknown pregnancy status:
  * P. falciparum cases: artemether-lumefantrine (AL) plus single dose primaquine (PQ) (0.25mg/kg daily)
  * P. vivax cases: chloroquine (CQ) plus 14 days of PQ (0.25mg/kg daily)
  * Mixed infections: AL plus 14 days of PQ (0.25mg/kg daily)
  Treatment for pregnant women and women breastfeeding children <6 months of age:
  * P. falciparum cases or mixed infections: Quinine (1st trimester); AL (2nd & 3rd trimesters or breastfeeding)
  * P. vivax cases: Chloroquine (CQ)
  Arms: Reactive Case Detection (RCD) arm
Other: Presumptive treatment with artemether-lumefantrine (AL) plus 14 days of primaquine (PQ) — Everyone who is eligible for the study except pregnant women and women breastfeeding children <6 months of age AND who are confirmed to have normal G6PD status will be treated presumptively with artemether-lumefantrine (AL) plus 14 days of primaquine (PQ). Treatment will be given without RDT for malaria.
  * Women in the first trimester of pregnancy will be treated presumptively with quinine.
  * Women in the second and third trimesters or women who are breastfeeding will receive artemether-lumefantrine (AL).
  Again, treatment will be given without RDT for malaria.
  Arms: Targeted Mass Drug Administration (tMDA) arm
Other: Optimized malaria control interventions — Optimized malaria control interventions that includes strengthened surveillance systems and commodities management, scale-up of vector control and case management services including follow-up, and social and behavior change communication to seek prompt treatment and use long lasting insecticidal nets (LLINs). Case management includes passive detection of malaria cases and treatment with artemether-lumefantrine (AL) plus single low dose primaquine (PQ) (0.25mg/kg once) for Plasmodium falciparum (Pf) cases and chloroquine (CQ) plus 14 days of PQ (0.25mg/kg daily) for Plasmodium vivax (Pv) cases, and AL plus 14 days of PQ (0.25mg/kg daily) for mixed infections as well as follow-up at the health post or health center on days 3, 7, and 13 for those receiving 14 days of PQ to assess for adverse events and adherence as per the national treatment guidelines.

SUMMARY:
Reactive and proactive case detection measures are widely implemented by national malaria elimination programs globally. Similarly, the Ethiopian Federal Ministry of Health decided to include reactive case detection (RCD) and targeted mass drug administration (tMDA) approaches as part of their elimination strategy, along with rigorous evaluation. This study aims to evaluate the impact on annual parasite incidence (API) and cost-effectiveness of implementing tMDA and RCD within a 100-meter radius of passively detected index case, compared with standard of care in the control arm. In addition, cross-sectional surveys will measure the change in malaria prevalence over the two-year study intervention period. The aim is to generate evidence to inform Ethiopia's national strategy for malaria elimination.

DETAILED DESCRIPTION:
Study design: Cluster randomized controlled trial

Primary aim: To compare the effect of targeted mass drug administration (tMDA) versus reactive case detection (RCD) on reducing malaria incidence

Study site: Elimination targeted areas within East Hararghe Zones, Oromia Regional State, which is comprised of 24 woredas/districts

Cluster or unit of randomization: Kebeles will be randomized to the control, RCD or tMDA arms using simple randomization

Evaluation methods: The primary outcome measure of annual parasite incidence (API) will be obtained through routine surveillance data at all health facilities (health centers and health posts).

Secondary outcomes will be measured through cross-sectional surveys and study monitoring data:

1. Case investigation. At the time of diagnosis of the index case and enrollment of community members to the study, a short questionnaire will be administered to collect demographic data and assess malaria risk, including past malaria treatment and travel history, access to malaria interventions, occupation, etc.
2. Cross-sectional surveys. At baseline and end of the study period (year 2), cross-sectional household surveys will be conducted to assess malaria prevalence, household and individual risk factors for malaria, including access to malaria interventions. It will also assess knowledge of, attitude towards, and participation in the study intervention.
3. Longitudinal feasibility measurements: Coverage of RCD or tMDA in the target population, acceptability of RCD or tMDA in the target population, serious adverse event (SAE) reports, adherence measured by self-report and pill count, and cost data from all arms
4. Laboratory testing: The conventional rapid diagnostic test (RDT) for malaria will be used in the RCD arm. Dried blood spots (DBS) will be collected for molecular and serological testing during the cross-sectional surveys in all arms. DBS collected in incident cases as part of routine surveillance as well as during the RCD activities will also be utilized for antigen, antibody, and molecular testing. G6PD testing will be used in the RCD and tMDA arm to guide primaquine (PQ) treatment.

Sample size: To measure the primary outcome, change in incidence, 16,000 Households (HH) (16 clusters, 1,000 HH each) per arm will be included in the study. For the cross-sectional surveys, 320 randomly selected HHs per arm (16 clusters, 20HH/cluster) will be included.

ELIGIBILITY:
Inclusion Criteria:

* Woreda-level: Of the 19 woredas with malaria risk, the ten woredas with the highest annual parasite incidence (API) in 2018 will be eligible for the study.
* For Kebeles:

  * Kebeles in East Hararghe Zone targeted for implementation of elimination activities by the Ethiopian Federal Ministry of Health where there is ongoing PMI-supported malaria surveillance;
  * Kebeles with reported API between 1 and 50;
  * Kebeles in malarious districts with comparable optimization of malaria control interventions.
* For individual participants:

  * All residents of the intervention study kebeles diagnosed with malaria at health facilities (index case) or reside within 100-meter radius with the index case and has NONE of the exclusion criteria listed below
  * Able to provide informed written consent

Exclusion Criteria:

* For kebeles: Kebeles planning on starting for the first time or discontinuing indoor residual spraying (IRS) campaigns in the next two years.
* For individual participants:

  * Children less than 6 months of age or <5 kg
  * Known allergy or history of adverse reaction or chronic/congenital disease contra indicated to any of the intervention drugs: PQ, AL or CQ
  * Individuals with severe malnutrition or signs of severe disease, with evidence of any organ failure or Hgb level < 8gm/dl
  * Household members already covered by the intervention less or equal to one month before

In addition, the following individuals will be excluded from receiving primaquine:

* Phenotypically G6PD deficient individuals
* Pregnant women
* Lactating women breastfeeding infants less than 6 months of age or with unknown G6PD status

Min Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 48960 (Estimated)
Dates: Start 2020-01-20 (Actual); Primary Completion 2022-01-20 (Estimated); Study Completion 2022-01-20 (Estimated)

PRIMARY OUTCOMES:
Change in malaria annual parasite incidence (API) | Two years
  The effect of RCD or tMDA will be defined as a change in malaria API among residents measured by microscopy/RDT through health centers and health posts. The malaria API will be defined as all passively detected RDT or microscopy confirmed cases over a period of 12 months, who are residents of the kebele divided by the estimated population in the intervention kebele multiplied by 1000. The primary effectiveness endpoint will therefore be API among residents of the kebele at baseline and year 2 of each intervention group of study clusters, compared with the control clusters.

SECONDARY OUTCOMES:
Malaria burden, measured by antigen test | Two years
  Testing for pan-Plasmodium antigens aldolase and LDH will determine active infection with malaria parasite, and, if the infecting species is Pf, by the presence of HRP2 antigen (Plucinski, Herman et al. 2018).
Malaria burden, measured by serology | Two years
  Sero-prevalence will be determined using LUMINEX based multiplex assays. Age-specific sero-conversion and sero-reversion rates over the two years will be used to monitor changes in transmission and malaria exposure over time. Absence of antimalarial antibodies, particularly in children, will show the success of tMDA or RCD interventions. Antigen selection will be informed by recent studies by EPHI and CDC and a panel of antibodies characterized to indicate recent change in transmission will be included (Kerkhof, Sluydts et al. 2016).
Malaria burden, measured by molecular testing | Two years
  Real-time quantitative (qPCR) for parasite detection will be performed by targeting the 18S small rRNA gene for Pf and Pv using primer and probe sequences. Pf parasites will be quantified using standard curves generated from a serial dilution of NF54 ring stage parasites. Pv parasite quantification will be done using plasmid constructs to infer copy numbers as described before. Blood samples in RNA protect buffers will be used for extraction of RNA using the RNeasy Mini Kit (QIAGEN) for gametocyte quantification, gametocyte commitment and maturation assays, sex ratio estimation, asexual stage parasites detection, and expression level of regulators of the balance between reproduction and replication.
Intervention coverage | Two years
  To compare intervention coverage in RCD and tMDA arms. After RCD and tMDA interventions, coverage will be estimated by calculating the proportion of all enumerated household members reached in each index case event and the proportion of individuals tested and/or on treatment.
Acceptability | Two years
  To compare acceptability of RCD and tMDA. During the baseline and endline cross-sectional surveys, the household head will be asked questions about the acceptability of the RCD and tMDA interventions (self-report).
Serious adverse events | Two years
  To compare number of serious adverse events between the RCD and tMDA arms
Adherence | Two years
  To compare the adherence to antimalarials between the RCD and tMDA arms. Adherence will be measured by self-report and pill count.
Costs | Two years
  To compare the costs of RCD and tMDA. Costs will be calculated using an ingredients approach that involves enumerating both the quantity of specific inputs (e.g., hours spent, cost of treatment, number of RDTs used, etc.) and the time spent during the intervention. Quantity and time will be converted to a common monetary cost measure. Existing infrastructure and recurrent inputs that would be present in the absence of the intervention will not be included in cost analysis. The emphasis of the cost analysis is on determining the cost of RCD and tMDA alone.
Cost-effectiveness | Two years
  To assess the cost-effectiveness of RCD and tMDA relative to control. Cost-effectiveness will be measured through incident malaria cases averted as measured through the difference in malaria incidence in RCD and tMDA kebeles.
Sensitivity and specificity of polymerase chain reaction (PCR) | Two years
  To evaluate the sensitivity and specificity of PCR as compared to antigen- based multiplex testing
Ratio of imported to locally acquired incident cases | Two years
  To assess the ratio of imported to locally acquired incident cases

CONTACTS AND LOCATIONS:
Overall Officials: Endalamaw Gadisa, PhD, MSc, Principal Investigator — AHRI Ethiopia
Locations (10):
- Ethiopia (10):
  - Woreda 1:, Babīlē
  - Woreda 2:, Fedīs
  - Woreda 3:, Girawa
  - Woreda 4:, Golo Oda
  - Woreda 5:, Gursum
  - Woreda 7:, Kersa
  - Woreda 8:, Kombolcha
  - Woreda 9:, Kurfa Chele
  - Woreda 10:, Midega Tola
  - Woreda 6:, ‘Alemaya

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Abdelmenan S, Teka H, Hwang J, Girma S, Chibsa S, Tongren E, Murphy M, Haile M, Dillu D, Kassim J, Behaksra S, Tadesse FG, Yukich J, Berhane Y, Worku A, Keating J, Zewde A, Gadisa E. Evaluation of the effect of targeted Mass Drug Administration and Reactive Case Detection on malaria transmission and elimination in Eastern Hararghe zone, Oromia, Ethiopia: a cluster randomized control trial. Trials. 2022 Apr 7;23(1):267. doi: 10.1186/s13063-022-06199-8. PMID 35392979

DOCUMENTS (1):
  • Informed Consent Form (2019-07-03): https://cdn.clinicaltrials.gov/large-docs/05/NCT04241705/ICF_000.pdf